CLINICAL TRIAL: NCT01811693
Title: The Field Administration of Stroke Therapy-Blood Pressure Lowering Pilot Trial
Brief Title: Field Administration of Stroke Therapy-Blood Pressure Lowering
Acronym: FAST-BP
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The funding period for the study has ended.
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Jeffrey L. Saver, Principal Investigator, University of California, Los Angeles
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FBP001
Record Dates: First submitted 2013-03-06; First posted 2013-03-14 (Estimated); Results first posted 2020-10-29 (Actual); Last update posted 2020-10-29 (Actual); Status verified 2020-10

CONDITIONS: Intracerebral Hemorrhage; Ischemic Stroke
Keywords: Stroke; Intracerebral Hemorrhage; Prehospital; Antihypertensive
MeSH Terms: conditions — Cerebral Hemorrhage; Ischemic Stroke; Stroke | interventions — Nitroglycerin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Dose Tier 1 (Experimental): Glycerly Trinitrate (Nitroglycerine) 5mg/24hour (0.2mg/hour) transdermal
  Interventions: Drug: Glycerly Trinitrate
- Dose Tier 2 (Experimental): Glycerly Trinitrate (Nitroglycerine) 10mg/24hour (0.4mg/hour) transdermal
  Interventions: Drug: Glycerly Trinitrate
- Dose Tier 3 (Experimental): Glycerly Trinitrate (GTN, Nitroglycerine) 5mg/24hour (0.2mg/hour) transdermal plus a single metered dose 0.4mg of sublingual GTN
  Interventions: Drug: Glycerly Trinitrate

INTERVENTIONS:
Drug: Glycerly Trinitrate — 5mg/24hour (0.2mg/hour) transdermal
  Other Names: Nitroglycerine; GTN
  Arms: Dose Tier 1
Drug: Glycerly Trinitrate — 10mg/24hour (0.4mg/hour) transdermal
  Other Names: Nitroglycerine; GTN
  Arms: Dose Tier 2; Dose Tier 3
Drug: Glycerly Trinitrate — 0.4 mg sublingual single metered spray
  Other Names: Nitroglycerine; GTN
  Arms: Dose Tier 3

SUMMARY:
This is an open, pilot, dose-escalation study of glyceryl trinitrate (GTN, Nitroglycerin) administered by paramedics in the field within 2 hours of symptom onset to 45 severely hypertensive stroke patients. The primary objective of the study is to evaluate the feasibility, safety, and physiologic efficacy of field-initiated glyceryl trinitrate in achieving modest reduction of blood pressure. Patients with acute stroke will be identified in the field by paramedics who have received training in basic and advanced cardiac life support, stroke recognition, and specific procedures relevant to the proposed study. Physician-investigators will obtain informed consent for each subject for study entry after cellular phone contact with paramedics. Paramedics will initiate antihypertensive treatment by applying transdermal GTN patch in the first two dose-tiers, and administering a single sublingual GTN metered spray followed by application of the transdermal system in the last dose tier. The sites involved in the study will be emergency medical services rescue ambulances and 8 receiving Stroke Center hospitals in Orange County, California, USA.

DETAILED DESCRIPTION:
The central aim of this phase 2a study is to identify a regimen of paramedic initiated glyceryl trinitrate antihypertensive therapy in acute stroke patients that is safe, is technically effective in modestly lowering blood pressure, and is optimal to advance to a pivotal trial. The study design is an open-label dose escalation study with three dose tiers,. It is anticipated that the trial will identify the most promising prehospital GTN regimen to advance to a pivotal, placebo-controlled, phase 3 trial.

Primary Hypothesis: Prehospital glyceryl trinitrate treatment reduces severely hypertensive blood pressure elevation by ED arrival.

The primary study endpoint to test this hypothesis will be the mean change in SBP from pre-treatment to ED arrival.

Secondary Hypotheses:

1. Prehospital glyceryl trinitrate treatment reduces severely hypertensive blood pressure elevation at early post-arrival timepoints and increases the proportion of patients with target blood pressure at ED arrival and early post-arrival timepoints.

   The secondary study endpoints analyzed to test these hypotheses will be: 1) mean change in SBP from pre-treatment to 30 minutes after ED arrival and 60 minutes after ED arrival; and 2) the proportion of patients with SBP < 180 mm Hg at ED arrival, 30, and 60 minutes after arrival.
2. Prehospital initiation of glyceryl trinitrate in the first 2 hours for severely hypertensive patients with stroke is feasible and safe.

Safety of GTN in the first 2 hours for severely hypertensive stroke patients will be assessed by analysis of serious adverse events, neurologic change, and mortality. We hypothesize that initiation of treatment of the patients in the field will be associated with a favorable side effect profile and without severe blood pressure lowering to les than 120 mm Hg systolic.

Successful completion of the study will demonstrate feasibility to recruit hypertensive stroke participants and initiate GTN therapy in the field by paramedics.

ELIGIBILITY:
Inclusion Criteria:

1. Suspected stroke identified with Los Angeles Prehospital Stroke Screen
2. Age 40-80, inclusive
3. Last known well time within 2 hours of treatment initiation
4. Deficit present for > 15 minutes
5. Systolic blood pressure ≥180

Exclusion Criteria:

1. Coma
2. Rapidly improving neurologic deficit
3. Pre-existing neurologic, psychiatric, or advanced systemic disease that would confound the neurological or functional outcome evaluations
4. Severe respiratory distress (O2 sat < 90% or respiratory rate < 12 or > 24)
5. Major head trauma in the last 24 hours
6. Recent stroke within prior 30 days
7. Use of erectile dysfunction therapies in the previous 12 hours
8. Use of type V phosphodiesterase inhibitors
9. Patient unable to give informed consent and no available legally authorized representative (LAR) to provide informed consent

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2013-04; Primary Completion 2013-09-10 (Actual); Study Completion 2013-12-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Los Alamitos Medical Center, Los Alamitos, California
  - FAST-MAG Clinical Trial Coordinating Center, Los Angeles, California

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Dose Tier 1 | Dose Tier 2 | Dose Tier 3
Started | 4 | 0 | 0
Completed | 4 | 0 | 0
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The trial was stopped early due to slow enrollment. A pragmatic, low cost study, the lesser frequency of touchpoints between study staff and paramedics seemed to result in paramedics not reliably recalling in time that the study was available to offer to appropriate patients. Due to small sample size, some allocation cells had zero patients.
Groups:
- Total: Total of all reporting groups
Arm/Group | Dose Tier 1 | Dose Tier 2 | Dose Tier 3 | Total
Number analyzed (Participants) | 4 | 0 | 0 | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 0 | 0 | 2
  >=65 years | 2 | 0 | 0 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 0 | 2
  Male | 2 | 0 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Participants With Systolic Blood Pressure Change of 8mmHg or More
Description: The mean change in blood pressure was measured in the Emergency Department approximately 15 minutes after application of the treatment
Time Frame: Baseline, 15 minutes after treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Tier 1
Number analyzed (Participants) | 4
Participants | 1

2. Other Pre Specified Outcome: Participants Experiencing Serious Adverse Events
Time Frame: 90 days after enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Tier 1
Number analyzed (Participants) | 4
Participants
  SAE | 2
  No SAE | 2

3. Other Pre Specified Outcome: Participants Exhibiting Neurological Deterioration as Indicated by a Two-point or Greater Worsening in the Glasgow Coma Scale
Description: The Glasgow Coma Scale (GCS) score measures level of consciousness in eye, motor, and verbal components. At least one point is given in each category. The scale ranges from 3 to 15, with 3 indicating deep unconsciousness and 15 indicating consciousness is not impaired.
Time Frame: Baseline, One hour after enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Tier 1
Number analyzed (Participants) | 4
Participants | 1

4. Other Pre Specified Outcome: Participants With Systolic Blood Pressure Less Than 120 mm/Hg
Time Frame: 24 hours after enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Tier 1
Number analyzed (Participants) | 4
Participants | 0

ADVERSE EVENTS:
Time Frame: 90 days after enrollment
Arm/Group | Dose Tier 1
Serious Adverse Events (participants affected / at risk) | 2/4
Other Adverse Events (participants affected / at risk) | 0/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Tier 1 (N=4)
Death (Vascular disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No